CLINICAL TRIAL: NCT03454048
Title: Controlled Human Malaria Infection Study to Assess Gametocytemia and Mosquito Transmissibility in Participants Challenged With Plasmodium Falciparum by Sporozoite or Blood Stage Challenge to Establish a Model for the Evaluation of Transmission-blocking Interventions
Brief Title: Controlled Human Malaria Infection Model for Evaluation of Transmission-blocking Interventions - Study 2
Acronym: CHMI-trans2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other); QIMR Berghofer Medical Research Institute (Other)
Responsible Party: Principal Investigator, Robert Sauerwein, Prof. dr., Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHMI-trans2
Record Dates: First submitted 2018-02-27; First posted 2018-03-05 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-03

CONDITIONS: Malaria,Falciparum; Gametocytes; Controlled Human Malaria Infection; Transmission
MeSH Terms: conditions — Malaria, Falciparum | interventions — piperaquine; fanasil, pyrimethamine drug combination; atovaquone, proguanil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP (Experimental): Cohort A will be subjected to a standard controlled human malaria infection (CHMI) delivered by five Pf-infected mosquitoes. All volunteers will be treated with a single oral subcurative low-dose of piperaquine (LD-PIP, 480 mg, T1). Volunteers will receive a second treatment (T2, LD-PIP2, 480mg) if a recrudescence of asexual parasitemia occurs before day 21 post challenge infection. Volunteers in group 1 (LD-PIP/LD-PIP2/PIP) will be curatively treated with piperaquine (960mg).
  Interventions: Drug: Piperaquine (low dose); Drug: Piperaquine (high dose); Drug: Atovaquone Proguanil; Other: malaria challenge infection, P. falciparum 3D7
- Group 2 (Cohort A) LD-PIP/LD-PIP2/SP (Experimental): Cohort A will be subjected to a standard controlled human malaria infection (CHMI) delivered by five Pf-infected mosquitoes. All volunteers will be treated with a single oral subcurative low-dose of piperaquine (LD-PIP, 480 mg, T1). Volunteers will receive a second treatment (T2, LD-PIP2, 480mg) if a recrudescence of asexual parasitemia occurs before day 21 post challenge infection. Volunteers in group 2(LD-PIP/LD-PIP2/SP) will be curatively treated with sulfadoxine-pyrimethamine (1000mg/50mg).
  Interventions: Drug: Piperaquine (low dose); Drug: Sulfadoxine pyrimethamine; Drug: Atovaquone Proguanil; Other: malaria challenge infection, P. falciparum 3D7
- Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP (Experimental): Cohort B will be subjected to a standard blood stage challenge with ~2,800 Pf-infected erythrocytes by intravenous injection. All volunteers will be treated with a single oral subcurative low-dose of piperaquine (LD-PIP, 480 mg, T1). Volunteers will receive a second treatment (T2, LD-PIP2, 480mg) if a recrudescence of asexual parasitemia occurs before day 21 post challenge infection. Volunteers in group 3 (LD-PIP/LD-PIP2/PIP) will be curatively treated with piperaquine (960mg)
  Interventions: Drug: Piperaquine (low dose); Drug: Piperaquine (high dose); Drug: Atovaquone Proguanil; Other: Blood stage malaria challenge infection, P. falciparum 3D7
- Group 4 (Cohort B) LD-PIP/LD-PIP2/SP (Experimental): Cohort B will be subjected to a standard blood stage challenge with ~2,800 Pf-infected erythrocytes by intravenous injection. All volunteers will be treated with a single oral subcurative low-dose of piperaquine (LD-PIP, 480 mg, T1). Volunteers will receive a second treatment (T2, LD-PIP2, 480mg) if a recrudescence of asexual parasitemia occurs before day 21 post challenge infection. Volunteers in group 4 (LD-PIP/LD-PIP2/SP) will be curatively treated with sulfadoxine-pyrimethamine (1000mg/50mg).
  Interventions: Drug: Piperaquine (low dose); Drug: Sulfadoxine pyrimethamine; Drug: Atovaquone Proguanil; Other: Blood stage malaria challenge infection, P. falciparum 3D7

INTERVENTIONS:
Drug: Piperaquine (low dose) — subcurative regimen (480 mg)
  Other Names: piperaquine phosphate
Drug: Piperaquine (high dose) — Curative regimen (960mg)
  Other Names: piperaquine phosphate
  Arms: Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP; Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP
Drug: Sulfadoxine pyrimethamine — Curative regimen (1000mg/50mg)
  Other Names: Fansidar
  Arms: Group 2 (Cohort A) LD-PIP/LD-PIP2/SP; Group 4 (Cohort B) LD-PIP/LD-PIP2/SP
Drug: Atovaquone Proguanil — Curative regimen (1000/400 mg, for 3 days)
  Other Names: Malarone
Other: malaria challenge infection, P. falciparum 3D7 — malaria challenge infection by P. falciparum 3D7-infected mosquito bites
  Other Names: 3D7 Plasmodium falciparum
  Arms: Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP; Group 2 (Cohort A) LD-PIP/LD-PIP2/SP
Other: Blood stage malaria challenge infection, P. falciparum 3D7 — P. falciparum 3D7-infected human erythrocytes administered intravenously for the purpose controlled human malaria infection.
  Other Names: P. falciparum 3D7-infected human erythrocytes
  Arms: Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP; Group 4 (Cohort B) LD-PIP/LD-PIP2/SP

SUMMARY:
This is a single-center, open label study. The primary aim of this project is to develop a controlled human malaria infection transmission model ("CHMI-trans") or "challenge model" to evaluate the capacity of vaccines, biologics (monoclonal antibodies, or mAbs), and drugs to block malaria parasite transmission by assessing infectiousness of Plasmodium falciparum (Pf) gametocyte carriers for Anopheles mosquitoes.

DETAILED DESCRIPTION:
A total of 24 volunteers, in two cohorts (n=12), will be randomly assigned to two groups per cohort (n=6). Cohort A will be subjected to a standard controlled human malaria infection (CHMI) delivered by five Pf-infected mosquitoes (groups 1 and 2). Cohort B will be subjected to a standard blood stage challenge with ~2,800 Pf-infected erythrocytes by intravenous injection (groups 3 and 4).

Treatment is subsequently initiated to induce gametocytemia (treatment 1, T1) and to clear pathogenic asexual parasites whilst leaving gametocytes unaffected (treatment 2 and 3, T2 and T3). At the end of the study, treatment of all parasite stages is provided following national treatment guidelines (end treatment, ET).

Once malaria infections are detected by 18S qPCR positive (sporozoite challenge) or on day 8 (blood stage challenge), all volunteers will be treated with a single oral subcurative low-dose of piperaquine (LD-PIP, 480 mg, T1). Using blood samples taken twice daily, the initial clearance of parasitemia will be carefully monitored. After T1, volunteers will receive a second treatment (T2, LD-PIP2, 480mg) if a recrudescence of asexual parasitemia occurs before day 21 post challenge infection. On day 21 or when a recrudescence occurs after T2, volunteers in group 1 and 3 (LD-PIP/LD-PIP2/PIP) will be curatively treated with piperaquine (960mg) and group 2 and 4 (LD-PIP/LD-PIP2/SP) with sulfadoxine-pyrimethamine (1000mg/50mg). These treatment regimens cure asexual parasitemia while leaving immature and mature gametocytes unaffected. To ensure the radical clearance of all parasite stages, all volunteers will receive a final treatment (ET) according to national guidelines with atovaquone/proguanil (Malarone®) on day 36. Daily blood samples will allow detailed quantification of gametocytes, gametocyte sex ratio and ex vivo assessments of gametocyte fitness. Additionally, blood samples will be obtained for Direct Membrane Feeding Assay (DMFA) and volunteers will be subjected to Direct Skin Feeding Assays (DFA). These assays will provide evidence on the infectivity of volunteers.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Subject is aged ≥ 18 and ≤ 35 years and in good health.
2. Subject has adequate understanding of the procedures of the study and is able and willing (in the investigator's opinion) to comply with all study requirements.
3. Subject is willing to complete an informed consent questionnaire and is able to answer all questions correctly.
4. Subject is able to communicate well with the investigator and is available to attend all study visits, lives in proximity to the trial centre (<10 km) or (if >10km) is willing to stay in a hotel close to the trial centre during part of the study (from day 4 (blood stage challenge) 5 (sporozoite challenge) post-infection until T1+4 provided that the subject has had 2 consecutive negative 18S qPCR tests (at least 24 hours apart) following T1 treatment; or until day T3+3).
5. The subject will remain within the Netherlands during the challenge period, will not travel to a malaria-endemic area during the study period, and is reachable (24/7) by mobile telephone throughout the entire study period.
6. Subject agrees to their general practitioner being informed and contacted about their participation in the study and agrees to sign a form to request the release by their General Practitioner (GP), and medical specialist when necessary, to the investigator(s), of any relevant medical information concerning possible contra-indications for participation in the study.
7. The subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period and for a defined period thereafter according to current Sanquin guidelines.
8. For female subjects: subject agrees to use continuous adequate contraception** and not to breastfeed for the duration of study.
9. Subject agrees to refrain from intensive physical exercise (disproportionate to the subject's usual daily activity or exercise routine) during the malaria challenge period until day 38 after infection.
10. Subject agrees to avoid additional triggers that may cause elevations in liver enzymes including alcohol from baseline up to 1 week post treatment (T3).
11. Subject has signed written informed consent to participate in the trial. (*Acceptable forms of contraception include: established use of oral, injected or implanted hormonal contraceptives; intrauterine device or intrauterine system; barrier methods (condoms or diaphragm with additional spermicide); male partner's sterilisation (with appropriate post-vasectomy documentation of absence of sperm in the ejaculate); true abstinence when this is in line with the preferred and usual lifestyle of the subject; Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immunodeficient, psychiatric and other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following.

   1.1. Body weight <50 kg or Body Mass Index (BMI) <18 or >30 kg/m2 at screening. 1.2. A heightened risk of cardiovascular disease, as determined by: an estimated ten year risk of fatal cardiovascular disease of ≥5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE); history, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities; or a positive family history of cardiac events in 1st or 2nd degree relatives <50 years old.

   1.3. A medical history of functional asplenia, sickle cell trait/disease, thalassaemia trait/disease or G6PD-deficiency.

   1.4. History of epilepsy in the period of five years prior to study onset, even if no longer on medication.

   1.5. Screening tests positive for Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) 1.6. Chronic use of i) immunosuppressive drugs, ii) antibiotics, iii) or other immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period.

   1.7. Any recent or current systemic therapy with an antibiotic or drug with potential anti-malarial activity (chloroquine, doxycycline, tetracycline, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, erythromycin, hydroxychloroquine, etc.) (allowable timeframe for use at the Investigator's discretion).

   1.8. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years.

   1.9. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year.

   1.10. History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening or at inclusion, or positive urine toxicology test for cannabis at inclusion.
2. For female subjects: positive urine pregnancy test at screening and/or at the baseline visit.
3. Abnormal ALT/AST values on baseline
4. Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study.
5. Known hypersensitivity to or contra-indications (including co-medication) for use of sulfadoxine-pyrimethamine, piperaquine, chloroquine, Malarone®, artemether-lumefantrine, primaquine or history of severe (allergic) reactions to mosquito bites.
6. Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
7. Being an employee or student of the department of Medical Microbiology of the Radboudumc or the department of Internal Medicine.
8. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
9. For cohort B (blood stage challenge): Received a blood transfusion in the past.
10. For cohort B (blood stage challenge): Women of childbearing potential with a screening test positive for erythrocyte anti-Rh(c) and/or anti-Rh(e) antibodies.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Result] Alkema M, Reuling IJ, de Jong GM, Lanke K, Coffeng LE, van Gemert GJ, van de Vegte-Bolmer M, de Mast Q, van Crevel R, Ivinson K, Ockenhouse CF, McCarthy JS, Sauerwein R, Collins KA, Bousema T. A Randomized Clinical Trial to Compare Plasmodium falciparum Gametocytemia and Infectivity After Blood-Stage or Mosquito Bite-Induced Controlled Malaria Infection. J Infect Dis. 2021 Oct 13;224(7):1257-1265. doi: 10.1093/infdis/jiaa157. PMID 32239171

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP | Group 2 (Cohort A) LD-PIP/LD-PIP2/SP | Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP | Group 4 (Cohort B) LD-PIP/LD-PIP2/SP
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP | Group 2 (Cohort A) LD-PIP/LD-PIP2/SP | Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP | Group 4 (Cohort B) LD-PIP/LD-PIP2/SP | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Median (Full Range); unit: years] | 24.5 [18 to 30] | 22.5 [19 to 26] | 25.5 [20 to 29] | 20.0 [19 to 26] | 24 [18 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 4 | 15
  Male | 3 | 2 | 2 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4 | 5 | 5 | 6 | 20
  Other/unknown | 2 | 1 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Netherlands | 6 | 6 | 6 | 6 | 24
Hemoglobin [Median (Full Range); unit: mmol/L] | 8.8 [8.0 to 9.7] | 8.2 [7.6 to 9.9] | 8.8 [7.6 to 10.0] | 8.7 [7.5 to 9.4] | 8.7 [7.5 to 10.0]
Body Mass Index (kg/m2) [Median (Full Range); unit: Kg/m^2] | 22.2 [20.8 to 29.3] | 24.2 [22.7 to 26.9] | 20.4 [18.1 to 22.8] | 24.7 [20.8 to 27.7] | 22.75 [18.10 to 29.3]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events in the CHMI-trans Model
Description: Frequency of adverse events in the CHMI-trans model.
Time Frame: up to day 51 after challenge infection
Measure: Number; unit: Adverse events
Arm/Group | Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP | Group 2 (Cohort A) LD-PIP/LD-PIP2/SP | Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP | Group 4 (Cohort B) LD-PIP/LD-PIP2/SP
Number analyzed (Participants) | 6 | 6 | 6 | 6
Adverse events | 95 | 95 | 107 | 52

2. Primary Outcome: Gametocyte Prevalence
Description: Number of individuals in each study arm that show prevalence of gametocytes as defined by quantitative reverse-transcriptase PCR (qRT-PCR) for CCp4 (female) and PfMGET (male) mRNA with a threshold of 5 gametocytes/mL for positivity.
Time Frame: up to day 51 after challenge infection
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP | Group 2 (Cohort A) LD-PIP/LD-PIP2/SP | Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP | Group 4 (Cohort B) LD-PIP/LD-PIP2/SP
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 5 | 6 | 6 | 6

3. Primary Outcome: Magnitude of Adverse Events in the CHMI-trans Model
Description: symptoms will be ranked as (1) mild, (2) moderate, or (3) severe, depending on their intensity according to the following scale:
  * Mild (grade 1): awareness of symptoms that are easily tolerated and do not interfere with usual daily activity
  * Moderate (grade 2): discomfort that interferes with or limits usual daily activity
  * Severe (grade 3): disabling, with subsequent inability to perform usual daily activity, resulting in absence or required bed rest
Time Frame: up to day 51 after challenge infection
Measure: Number; unit: Adverse events
Arm/Group | Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP | Group 2 (Cohort A) LD-PIP/LD-PIP2/SP | Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP | Group 4 (Cohort B) LD-PIP/LD-PIP2/SP
Number analyzed (Participants) | 6 | 6 | 6 | 6
Adverse events
  Mild (grade I) | 64 | 56 | 86 | 41
  Moderate (grade II) | 22 | 22 | 17 | 8
  Severe (grade III) | 9 | 17 | 4 | 3

4. Secondary Outcome: Peak Density Gametocytes
Description: Peak density of gametocytes by qRT-PCR.
Time Frame: up to day 51 after challenge infection
Measure: Median (Full Range); unit: Gametocytes/mL
Arm/Group | Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP | Group 2 (Cohort A) LD-PIP/LD-PIP2/SP | Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP | Group 4 (Cohort B) LD-PIP/LD-PIP2/SP
Number analyzed (Participants) | 6 | 6 | 6 | 6
Gametocytes/mL | 13.9 [2.5 to 727.9] | 21.4 [6.16 to 181.6] | 1442.2 [246.6 to 3826.1] | 813.2 [179.5 to 1617.0]

5. Secondary Outcome: AUC Gametocytes
Description: The area under the curve of gametocyte density versus time. The median AUC was calculated for both cohorts. Since onset of gametocytaemia differs depending on method of infection a window of 15 days was used to calculate AUC, from the time-point where a minimum of 50% of participants within a cohort had detectable gametocytemia.
Time Frame: up to day 51 after challenge infection
Population: Data are represented per inoculation method (Cohort A; mosquito bite infection, Cohort B; induced blood stage malaria) and not per study arm (group 1-4) as this better reflects the effects of inoculation route on induction of transmissible gametocytaemia.
Measure: Median (Full Range); unit: (gametocytes*days)/mL
Groups:
- Cohort A: Group 1 and 2
- Cohort B: Group 3 and 4
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 12
(gametocytes*days)/mL | 99 [16.6 to 5330] | 11043 [1643 to 37326]

6. Secondary Outcome: Gametocyte Commitment
Description: The gametocyte commitment rate is estimated by dividing the peak gametocyte by the peak of asexual parasites.
Time Frame: up to day 51 after challenge infection
Population: as for outcome 5
Measure: Median (Full Range); unit: gametocytes/asexual parasite
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 12
gametocytes/asexual parasite | 0.0011 [0.0002 to 0.0141] | 0.0323 [0.0121 to 0.0891]

7. Secondary Outcome: Gametocyte Sex-ratio
Description: Proportion of male gametocytes
Time Frame: up to day 51 after challenge infection
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Proportion of male gametocytes
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 12
Proportion of male gametocytes | 0.20 [0.14 to 0.50] | 0.31 [0.22 to 0.51]

8. Secondary Outcome: Number of Participants Infectious for Mosquitoes Through DFA
Description: Prevalence of gametocyte infectiousness for Anopheles mosquitoes through Direct Feeding Assays (Direct Skin Feeding Assay, DFA).
Time Frame: up to day 51 after challenge infection
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 12
Participants | 0 | 9

ADVERSE EVENTS:
Time Frame: From inclusion until 51 days post infection
Arm/Group | Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP | Group 2 (Cohort A) LD-PIP/LD-PIP2/SP | Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP | Group 4 (Cohort B) LD-PIP/LD-PIP2/SP
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Cohort A) LD-PIP/LD-PIP2/PIP (N=6) | Group 2 (Cohort A) LD-PIP/LD-PIP2/SP (N=6) | Group 3 (Cohort B) LD-PIP/LD-PIP2/PIP (N=6) | Group 4 (Cohort B) LD-PIP/LD-PIP2/SP (N=6)
Fever (Infections and infestations) | 6 (16) | 6 (11) | 6 (13) | 3 (5)
Headache (Infections and infestations) | 6 (27) | 6 (26) | 6 (33) | 6 (20)
Nausea (Infections and infestations) | 5 (13) | 4 (12) | 6 (9) | 3 (6)
Malaise (Infections and infestations) | 4 (8) | 4 (15) | 1 (3) | 2 (2)
Myalgia (Infections and infestations) | 1 (1) | 5 (6) | 4 (7) | 4 (5)
Fatigue (Infections and infestations) | 4 (7) | 5 (13) | 5 (12) | 3 (6)
Chills (Infections and infestations) | 6 (13) | 1 (2) | 4 (7) | 1 (2)
Syncope (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Infections and infestations) | 0 (0) | 2 (2) | 5 (6) | 2 (2)
Decreased appetite (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (3) | 0 (0)
Dizziness (Infections and infestations) | 2 (5) | 1 (3) | 2 (8) | 2 (4)
Diarrhea (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Palpitations (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Arthralgia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nonspecific thoracic pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT03454048/Prot_SAP_000.pdf